CLINICAL TRIAL: NCT01001247
Title: A Phase I, Open Label, Randomized, 4-way Crossover Trial to Evaluate the Pharmacokinetics of TMC278 25mg and 50mg in the Presence of Omeprazole 20mg q.d., in Healthy Subjects
Brief Title: TMC278-TiDP6-C154: Evaluation of the Possible Influence of Omeprazole Intake - and the pH Increase in the Stomach Triggered by Omeprazole Intake - on the Blood Levels of TMC278 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Compound Development Team Leader, Tibotec Pharmaceuticals, Ireland
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016267
Record Dates: First submitted 2009-10-23; First posted 2009-10-26 (Estimated); Last update posted 2010-07-09 (Estimated); Status verified 2010-07

CONDITIONS: HIV Infections
Keywords: TMC278-TiDP6-C154; TMC278-C154; TMC278; Healthy volunteers; omeprazole; proton pump inhibitor; HIV
MeSH Terms: conditions — HIV Infections | interventions — Rilpivirine; Omeprazole

INTERVENTIONS:
Drug: TMC278; Omeprazole

SUMMARY:
The purpose of this study is to investigate the extent by which intake of 20 mg once daily (q.d.) omeprazole influences the levels of TMC278 in the blood after intake of 25 mg q.d.. This study also investigates - in case levels of TMC278 are reduced when co-administered with omeprazole - whether a double dose of TMC278 (50 mg q.d.) or a separation of intake of both drugs by 12 hours may circumvent a decrease of TMC278 levels in the blood below the clinical effective concentration. Omeprazole is prescribed to reduce the production of gastric acid. Since TMC278 requires gastric acid to be properly dissolved and taken up in the blood circulation, intake of omeprazole has an influence on the levels of TMC278 in the blood circulation. This effect has been revealed in a previously conducted clinical trial, using the combination of 150 mg TMC278 q.d. and 20 mg q.d. omeprazole. The currently proposed study will also further explore the relationship between the levels of TMC278 in the blood at several time points and the acidity of the stomach. Also the short-term safety and tolerability of co-administration of omeprazole 20 mg q.d. and TMC278 25 mg q.d. will be assessed.

DETAILED DESCRIPTION:
This is an open label study, which means that all parties including the study doctor, the healthy volunteer and the sponsor plus his designees will know at all times which treatment the volunteer is in. This is a 4-way cross over trial, which means that every volunteer will be sequentially subjected to 4 different treatments.There are 4 treatment sequences defined: ABCD, BDAC, CADB and DCBA. Treatment sessions are organized in such a way that between successive intakes of TMC278 a period of 14 days is respected. Treatment A is the reference, showing the levels of TMC278 in blood without any intake of omeprazole. These data points will be compared with blood levels of TMC278 when TMC278 is being administered 1.5 hours after intake of omeprazole (Treatment B) or with blood levels of TMC278 when being administered 12 hours after intake of omeprazole (Treatment C). Treatment B will be the comparator of Treatment D, in order to reveal whether doubling the dose of TMC278 (50 mg q.d. used in Treatment D) can circumvent the reduction of TMC278 levels when being co-administered with omeprazole, if applicable. In each session, an extensive investigation of the levels of TMC278 in the blood circulation is planned. Levels of TMC278 will be assessed at 16 different time points, i.e. before administration of TMC278, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours after intake of TMC278. During all treatments, the acidity in the stomach (called intragastric pH) will be monitored during a 24-hour period on the day of TMC278 intake. Standard Safety assessments (blood biochemistry and haematology, urine analysis, ECG, pulse rate and blood pressure) will be performed on Day1, 2 and 8 in Treatment A and on Day-5, 1, 2, 8 in Treatment B, C and D. Treatment A: 25mg TMC278 in the morning of Day1; Treatment B: 25mg TMC278 in the morning of Day1 and 20mg omeprazole in the morning from Day-5 through Day2 (7 days in total); Treatment C: same as treatment B, but omeprazole is taken in the evening; Treatment D: same as treatment B, but 50mg omeprazole is taken instead of 25mg. All intakes are oral. In Treatment B, C and D, the intake of omeprazole is witnessed by site staff on Days -5, -3, -2 and -1

ELIGIBILITY:
Inclusion Criteria:

* Smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day (or non-smoking) for at least 3 months prior to selection
* Weight as defined by a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* Informed Consent Form (ICF) signed voluntarily
* Able to comply with protocol requirements
* Healthy on the basis of a pretrial physical examination, medical history, the results of blood biochemistry and hematology tests, a urinalysis, vital signs, and a 12-lead electrocardiogram (ECG)

Exclusion Criteria:

* No positive testing for HIV-1 or -2
* females, except if menopausal for at least 2 years, or with total hysterectomy or bilateral tubal ligation (without repair surgery)
* No infection of Hepatitis A, B or C
* No currently active gastrointestinal, cardiovascular, neurologic, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory or infectious disease
* No history of clinically relevant heart rhythm disturbances
* No positive urine drug testing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Plasma levels of TMC278 assessed after co-administration of 20mg q.d. omeprazole taken either in the morning (1.5 h before TMC278) or in the evening (12 h before TMC278); assess 24h intragastric pH at days of intake of TMC278 | Plasma levels: Treatment A, B, C and D: Day1 (at 11 time points), Day2, 3, 4, 6 and 8 (all at 1 time point). Intragastric pH: Treatment A, B, C and D at Day1 (=day of intake TMC278).

SECONDARY OUTCOMES:
To evaluate the short-term safety and tolerability of co-administration of omeprazole with a single 25mg and 50mg dose of TMC278 | 13 weeks (this includes a treatment, washout and follow up period and is excluding screening period of maximum 21 days before first medication intake)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited